CLINICAL TRIAL: NCT05777252
Title: Effects of 16-Week Circuit Training on Spine Structure, Trunk Muscle Endurance, and Balance in Healthy Women
Brief Title: Effects of 16-Week Circuit Training in Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Erhan Seçer, Lecturer, Celal Bayar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CBU-FTR-ES-O1
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Healthy Women
Keywords: Health status; Exercise; Spine; Physical fitness; Women
MeSH Terms: conditions — Motor Activity | interventions — Circuit-Based Exercise

STUDY DESIGN:
Intervention Model Description: Prospective clinic study with a single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training Group (Experimental): Circuit training will be applied to the participants for a total of 16 weeks, with an average of 40 minutes a day, 3 days a week, taking into account the recommendations of the American College of Sports Medicine (ACSM).
  Interventions: Other: Circuit Training

INTERVENTIONS:
Other: Circuit Training — Warm-up and cool-down protocols will be applied before and after each CT, and each exercise will be performed as 15 repetitions and an average of 40 seconds of rest will be given between exercises. Also, the intensity of CT will be determined according to the Borg scale (between 11 and 14). CT will include 'mini squat', 'step up', 'sit ups', 'reverse sit ups', 'leg press', 'leg curl', 'leg extension', 'crunches', 'lunge', 'prone bridge', and 'side bridge' exercises.

SUMMARY:
The aim of this study is to investigate the effects of 16-week CT on spine structure, trunk muscle endurance, and balance in healthy women.

DETAILED DESCRIPTION:
Circuit training (CT) was developed by Morgan and Anderson in 1953, and is a type of training that includes various exercise stations arranged in a certain order. During CT, each participant performs 8 to 20 repetitions of exercise at each station, usually in less than a minute. Also, each participant moves from one training station to another with short rest periods or without breaks, and ends a training session by completing all stations. This training includes exercises performed with only body weight without the use of any equipment or with ancillary equipment such as elastic bands, free weights, and exercise devices, or a combination of both types of exercise.

It is seen that CT, which is a method frequently preferred by individuals of all ages all over the world to improve or maintain both physical performance, and health-related fitness, is gaining popularity due to its practicality and efficiency in recent years. Especially, it has become an important exercise option for individuals who have the problem of 'not having enough time for exercise' in daily life. The fact that the intensity can be adjusted according to the individual participant, that it includes both aerobic exercises and strengthening and endurance exercises for the trunk, upper and lower extremity muscles, and that it aims to improve both the musculoskeletal and cardiovascular systems of the participants is an important factor that increases the preferability of this training in all populations. Also, it is reported that the inclusion of various types of exercise in this exercise training greatly reduces the rate of participants dropping out of this type of training or ending it completely compared to other types of training. Lastly, the main feature of this exercise training, which allows individual interaction both among the participants and between the participants and the sports or health professionals who provides this training, is that it includes a combination of different types of exercises in order to improve both the musculoskeletal, and cardiovascular systems.

In the literature, it was seen that studies investigating the effects of CT on trunk muscle endurance included different populations. However, there were few studies investigating the effects of CT on endurance of trunk muscles in healthy women. Also, it was seen that there was not enough evidence in the current literature about the effects of CT on the spine structure in healthy women. Especially, a possible increase in endurance of trunk muscles after training may also positively affect spine structure via the kinetic chain. Lastly, it was concluded that studies investigating the effects of CT on balance mostly included patients with neurological disorders or the youth population. A possible positive effects on the spine structure via the kinetic chain may improve balance by increasing neuromuscular control in healthy women. This issue needs detailed investigation.

Therefore, the aim of this study was to investigate the effects of 16-week CT on spine structure, trunk muscle endurance, and balance in healthy women. Also, the investigators hypothesized that the 16-week CT would be positive effects on spine structure, trunk muscle endurance, and balance in healthy women.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in study
* not have any systemic, neurological, or rheumatological disease

Exclusion Criteria:

* history of malignancy
* participating in another exercise training during the study
* using any medication that could affect the outcome of the study
* being pregnant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Being women
Enrollment: 34 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Posture (°) | Sixteen week
  Posture will be assessed with the Spinal Mouse® (Switzerland) device. The device has a measurement option different planes, provides the opportunity to evaluate both the posture and mobility of the spine, and gives valid, and reliable results. During the assessment, the processus spinosus of the spine from C7 to S3 will be marked and the mouse will be slide along the spine from top to bottom from the skin surface at a constant speed and pressure. Assessment were performed in an upright position for spinal posture.
Mobility (°) | Sixteen week
  Mobility will be assessed with the Spinal Mouse® (Switzerland) device. The device has a measurement option different planes, provides the opportunity to evaluate both the posture and mobility of the spine, and gives valid, and reliable results. During the assessment, the processus spinosus of the spine from C7 to S3 will be marked and the mouse will be slide along the spine from top to bottom from the skin surface at a constant speed and pressure. The assessment were performed in maximum forward flexion position for spine mobility.
Postural Competency (°) | Sixteen week
  Mobility will be assessed with the Spinal Mouse® (Switzerland) device. The device has a measurement option different planes, provides the opportunity to evaluate both the posture and mobility of the spine, and gives valid, and reliable results. During the assessment, the processus spinosus of the spine from C7 to S3 will be marked and the mouse will be slide along the spine from top to bottom from the skin surface at a constant speed and pressure. The assessment were performed in raising stretched-out arms to shoulder height with weights, designed according to the body weight, in each hand for postural competency.

SECONDARY OUTCOMES:
Trunk Muscle Endurance (sec) | Sixteen week
  Trunk muscle endurance will be measured with the trunk muscle endurance tests namely trunk flexion and extension endurance tests. Participants will be explained how to perform the positions by demonstrating them in advance. Then, they will be asked to repeat these positions once and to recognize the evaluation positions. Participants will be encouraged to maintain isometric postures for each test position as long as possible. The length of time that participants could maintain the correct position was recorded in seconds. This test does not contain minimum and maximum values. The longer the participants can maintain the correct position, the higher the endurance.
Balance | sixteen week
  Static balance will be assessed with the Biodex Balance System (Biodex Medical Systems, Inc., Shirley, New York, USA), which is a valid and reliable method (device), while the eyes are open and closed (bilateral) positions. Measurements will be repeated three times for static mode on barefoot. During the evaluation, the participant will be asked to give equal weight to both lower extremities on the platform and to remain as balanced as possible. This system (device) does not contain minimum and maximum values. A low score will be obtained from the device after the assessment indicates that the participant's balance performance is good.

CONTACTS AND LOCATIONS:
Overall Officials: Derya Ozer Kaya, Principal Investigator — Izmir Katip Celebi University; Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (2):
- Turkey (Türkiye) (2):
  - Izmir Katip Celebi University, Izmir
  - İzmir Katip Celebi University, Izmir

IPD SHARING:
Plan to Share IPD: No
The investigators do not want to share individual participant data